CLINICAL TRIAL: NCT00413595
Title: Stroke in Young Fabry Patients (sifap2): Characterization of the Stroke Rehabilitation in Young Patients With Fabry Disease: An Epidemiological, International, Multicenter Prognosis Study
Brief Title: Stroke in Young Fabry Patients (sifap2): Characterization of the Stroke Rehabilitation
Acronym: sifap2
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Collaborators: Shire Human Genetic Therapies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: II PV04/2006
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2020-04

CONDITIONS: Fabry Disease; Cerebrovascular Accident
Keywords: Cerebrovascular Accident; Cerebrovascular Accident, Acute; Fabry Disease; Fabry's Disease; Anderson-Fabry Disease; CVA (Cerebrovascular Accident); Stroke, acute; Cerebral Stroke
MeSH Terms: conditions — Fabry Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA-blood and urine sample for central laboratory analysis of agalsidase antibodies and Gb3 for safety issues.
  There will be a proteomic analysis in blood to check whether there will be the possibility to characterize a biomarker for Fabry disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Adult patients (18 - 55 years of age) with an acute cerebrovascular event of any etiology and the genetic diagnosis (a-galactosidase defect) of Fabry disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational, epidemiological, prognosis study; no drug tested; only laboratory analysis and diagnostic interventions done.

SUMMARY:
New studies indicate that in about 1 - 2 percent of the younger stroke patients the cause could have been an undiagnosed genetic disease, the so called Fabry disease. In this case certain fat molecules are not digested and broken down by the body - but remain in the cells. These fat molecules build up to dangerous levels, which start to damage the body, because they accumulate e.g. in the walls of the blood vessels. This accumulation in the blood vessels of the whole body may cause life-threatening malfunctions in the brain, inducing a stroke.

The purpose of this study is to investigate the stroke rehabilitation of Fabry patients during different therapeutic standard approaches for stroke and for Fabry disease (if any). During this study, stroke patients with Fabry disease will be monitored in greater detail to determine whether the differences in treatment are significant for patient recovery and on what they depend.

DETAILED DESCRIPTION:
In a group of young stroke patients with diagnosed Fabry disease the stroke rehabilitation will be investigated during different prophylactic therapeutic approaches. In this study the investigator will not be given any instructions on stroke and Fabry therapy.

All patients with any etiology of stroke and a diagnosed Fabry disease submitted to the stroke unit of the participating centres which commit to work with the EUSI (European Stroke Initiative) recommendations for stroke management and diagnosis will be included into the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 - 55 years of age) with an acute cerebrovascular event (CVE) of any etiology defined as patients having an ischemic stroke or transient ischemic attack
* Genetic diagnosis (a-galactosidase defect)of Fabry disease
* Written informed consent from patient

Exclusion Criteria:

* No proven Fabry disease
* Participating in an other clinical trial with any investigational new drug or medical device
* Contraindication to any of the diagnostic procedures like e.g. MRI investigation
* Patient has been pretreated with Enzyme Replacement Therapy at the date of informed consent of sifap2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients (18 - 55 years of age) with an acute cerebrovascular event (CVE) of any etiology defined as patients having an ischemic stroke or transient ischemic attack and genetic diagnosis (a-galactosidase defect) of Fabry disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-07 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Determination of the relapse rate of acute cerebrovascular events with clinical relevance in patients with different prophylactic approaches | 54 months study duration

SECONDARY OUTCOMES:
Quality of Life measured with the SF-36 | 54 months study duration
Number of acute CVEs without clinical significance but with obvious signs in MRI diagnosis | 54 months study duration
Beck Depression Inventory II (BDI II) | 54 months study duration
Brief Pain Inventory (BPI) | 54 months study duration
Rostocker Kopfschmerzfragen-Komplex (RoKoKo) (only in Austria and Germany) | 54 months study period
Habi test (only in Austrian and German centers) | 54 months study duration
Trail Making Test (TMT) | 54 months study duration
Functional neurological deficits measured by the Mini Mental State Examination (MMSE) | 54 months study duration

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof., MD, Principal Investigator — University of Rostock, Albrecht-Kossel-Institute for Neuroregeneration
Locations (20):
- Universitätsklinikum für Neurologie, Graz, Austria
- Department of Neurology, University Hospital Sestre Milosrdnice, Zagreb, Croatia
- Hopital Neurologique de Lyon, Service d'urgences Neurovasculaires, Lyon, France
- Department of Neurology, S. Khechinashvili University clinic of Tbilisi state medical university, Tbilisi, Georgia
- Germany (14):
  - Department of Neurology, Klinikum Hohe Warte, Bayreuth
  - Charite Campus Benjamin Franklin, Dept. of Neurology, Berlin
  - Department of Neurology, Allgemeines Krankenhaus Celle, Celle
  - Department of Neurology, Klinikum Chemnitz gGmbH, Chemnitz
  - Department of Neurology, Universitaetsklinikum Carl Gustav Carus, Dresden
  - Heinrich-Heine-University Duesseldorf, Dept. of Neurology, Düsseldorf
  - University of Giessen-Marburg Dept. of Neurology, Giessen
  - Department of Neurology, Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Department of Neurology, Universitaetsklinikum Jena, Jena
  - Department of Neurology, Universitaetsklinikum Leipzig, Leipzig
  - Dept. of Neurology, Ökumenisches Hainich Klinikum gGmbH, Mühlhausen
  - Ludwig-Maximilians-University of Munich, Klinikum München-Großhadern, Dept. of Neurology, München
  - Department of Neurology, University Tuebingen, Tübingen
  - University of Ulm, Department of Neurology, Ulm
- Institute of Psychiatry and Neurology, Dept. of Neurology, Warsaw, Poland
- Centro Hospitalar de Lisboa Central, Servico de Neurologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rolfs A, Bottcher T, Zschiesche M, Morris P, Winchester B, Bauer P, Walter U, Mix E, Lohr M, Harzer K, Strauss U, Pahnke J, Grossmann A, Benecke R. Prevalence of Fabry disease in patients with cryptogenic stroke: a prospective study. Lancet. 2005 Nov 19;366(9499):1794-6. doi: 10.1016/S0140-6736(05)67635-0. PMID 16298216